CLINICAL TRIAL: NCT01199536
Title: Observational Study to Evaluate Helicobacter Pylori Eradication at the End of Routine Triple Eradication Therapy With Duodenal Ulcer Relapses Control.
Brief Title: Helicobacter Pylori Eradication Treatment in Patients With Duodenal Ulcers
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GRU-NEX-2009/1
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Duodenal Ulcer
Keywords: Helicobacter-positive duodenal ulcer
MeSH Terms: conditions — Duodenal Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for Hematology (whole blood) and Chemistry (serum), gasric mucosa biopsies taken during esophagogastroduodenoscopy (EGDS) in routine practice of Moscow Medical Academy n/a I.M. Sechenov, Moscow State Medical and Stomatological University, Central Clinical Hospital of Presidential Administration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with Helicobacter-positive duodenal ulcer

SUMMARY:
The Study purpose is to evaluate Helicobacter pylori susceptibility to Clarithromycin and to estimate eradication and healing rates of duodenal ulcer routine eradication therapy at the end of treatment and 52 weeks from the therapy start

ELIGIBILITY:
Inclusion Criteria:

* Active duodenal ulcer with duodenal ulcer exacerbation confirmed by endoscopic signs of duodenal ulcer disease (acute ulcer or scar deformity of the duodenal bulb) and anamnesis data.
* Helicobacter pylori positive diagnosis at entry by 13C-Urea Breath Test (UBT)
* Prescription of the standard 7-day eradication therapy including esomeprazole 20 mg bd, amoxicillin 1000 mg bd, clarithromycin 500 mg bd
* Written informed consent provided prior the start of participation in the study.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent
* Current complication of duodenal ulcer disease, e.g. perforation, bleeding or pyloric stenosis
* History of esophageal/gastric/duodenal surgery except of the patients underwent perforated ulcer closure or endoscopic hemostasis more than 6 months ago
* Contraindications to Esomeprazole, Amoxicillin or Clarythromycin including known or suspected hypersensitivity or allergy
* Treatment with Amoxicillin, Clarythromycin or Bismuth containing drugs one month prior to inclusion
* Two or more previous attempts to eradicate H. Pylori

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Eradication rate of H. pylori at the end routine triple eradication therapy | 1 year

SECONDARY OUTCOMES:
Recurrence rate of duodenal ulcer (in patients with ulcer defects in inclusion stage) | 2 years
Frequency of duodenal ulcer relapses | 2 years
  Frequency of duodenal ulcer relapses based on gastroscopy data and recurrence rate of H.Pylori infection based on breath test data after 52 weeks from the start of the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir T. Ivashkin, Principal Investigator — Head of Chair of Internal Diseases Propedeutics and Gastroenterology at MMA n/a I.M. Sechenov
Locations (1):
- Research Site, Moscow, Russia